CLINICAL TRIAL: NCT04745689
Title: A Phase II Multicenter, Open-Label, Single Arm Study to Determine the Efficacy, Safety and Tolerability of AZD2811 and Durvalumab Combination as Maintenance Therapy After Induction With Platinum-Based Chemotherapy Combined With Durvalumab, for the First-Line Treatment of Patients With Extensive Stage Small-Cell Lung Cancer
Brief Title: Study of AZD2811 + Durvalumab in ES-SCLC
Acronym: TAZMAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6132C00001; 2024-511887-10-00 (Registry Identifier: EU (CTIS)); 2020-004091-18 (EudraCT Number)
Record Dates: First submitted 2020-12-16; First posted 2021-02-09 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Small-Cell Lung Cancer
Keywords: Extensive Stage Small-Cell Lung Cancer; Carcinoma, Small Cell Lung; Oat Cell Carcinoma of Lung; Oat Cell Lung Cancer; Small Cell Cancer Of The Lung; Small Cell Lung Cancer; SCLC; ES-SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; AZD2811; Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD2811 + Durvalumab (Experimental): Induction:
  Durvalumab + Platinum Chemotherapy (Carboplatin or cisplatin & Etoposide)
  Maintenance:
  AZD2811 + Durvalumab
  Interventions: Drug: Durvalumab; Drug: AZD2811; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Durvalumab — IV infusions through induction phase.
  IV infusions through maintenance phase until PD or other discontinuation criteria.
  Other Names: Imfinzi
Drug: AZD2811 — IV infusions through maintenance phase until PD or other discontinuation criteria.
Drug: Carboplatin — IV infusions through induction phase if chosen by Investigator.
Drug: Cisplatin — IV infusions through induction phase if chosen by Investigator.
Drug: Etoposide — IV infusions through induction phase.

SUMMARY:
A Phase II Multicenter, Open-Label, Single Arm Study to Determine the Efficacy, Safety and Tolerability of AZD2811 and Durvalumab Combination as Maintenance Therapy After Induction with Platinum-Based Chemotherapy Combined with Durvalumab, for the First-Line Treatment of Patients with Extensive Stage Small-Cell Lung Cancer.

DETAILED DESCRIPTION:
Primary objective of this study is to evaluate the efficacy of AZD2811 and durvalumab in patients who have not progressed following induction therapy with platinum-based chemotherapy combined with durvalumab.

This is an open-label, single arm study. Patients will be treated in an induction phase with platinum-based induction therapy and durvalumab. At the end of this induction period, participants will be assessed for disease progression, per RECIST v1.1.

Participants who have not progressed per RECIST v1.1 at the end of the induction phase will roll over into the maintenance phase of the trial, where patients will commence AZD2811 and durvalumab combination.

Participants will be treated with AZD2811 and durvalumab as maintenance therapy until confirmed progressive disease, start of non-protocol defined anticancer therapy, unacceptable toxicity, or withdrawal of consent.

If study intervention is permanently discontinued, the participant will remain in the study to be evaluated for safety assessment, as well as for confirmed disease progression and for survival.

Targeted population are adult patients (aged ≥18 years) with histologically or cytologically documented extensive disease (American Joint Committee on Cancer Stage (7th edition) IV SCLC [T any, N any,M1 a/b]), or T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan. Patients must have WHO/ECOG performance status of 0 or 1.

Tumor assessments will be performed at Screening as baseline with follow-up every 6 weeks ± 1 week for the first 36 weeks, and then every 8 weeks ±1 week until confirmed objective disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of extensive stage SCLC (ES-SCLC)
* Participants must be considered suitable to receive an induction platinum-based chemotherapy regimen, combined with durvalumab, as first-line treatment for ES-SCLC
* No prior exposure to immune-mediated therapy
* Life expectancy ≥12 weeks at Day 1.
* ECOG 0 or 1 at enrolment.

Exclusion Criteria:

* Any history of radiotherapy to the chest prior to systemic therapy or planned consolidation chest radiation therapy
* Has a paraneoplastic syndrome (PNS) of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents) or has a clinical symptomatology suggesting worsening of PNS
* Active infection including tuberculosis, HIV, hepatitis B and C
* Active or prior documented autoimmune or inflammatory disorders
* Uncontrolled intercurrent illness, including but not limited to interstitial lung disease.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2026-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (9):
- Research Site, Grand Rapids, Michigan, United States
- Poland (3):
  - Research Site, Bydgoszcz
  - Research Site, Olsztyn
  - Research Site, Poznan
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Jinju
  - Research Site, Seoul
- Spain (2):
  - Research Site, Seville
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://vivli.org/

REFERENCES:
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6132C00001&attachmentIdentifier=f48272f5-c24d-4426-bb1e-d458dbedede4&fileName=D6132C00001_CSPv9.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6132C00001&attachmentIdentifier=c243277c-be7f-47ed-81d5-75e2156c8f6a&fileName=D6132C00001_SAP.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6132C00001&attachmentIdentifier=e4afd46d-a950-49a7-9351-3fd3449f6f1e&fileName=d6132c00001-CSR.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Induction: Durvalumab + Platinum Chemotherapy (Carboplatin or cisplatin & Etoposide)
  Maintenance:
  Durvalumab monotherapy
- AZD2811 + Durva: Induction: Durvalumab + Platinum Chemotherapy (Carboplatin or cisplatin & Etoposide)
  Maintenance: AZD2811 + Durvalumab
Period: Overall Study
Arm/Group | Standard of Care | AZD2811 + Durva
Started | 22 | 9
Entered Induction Phase | 22 | 9
Entered Maintenance Phase | 13 | 9
Completed | 0 | 0
Not Completed | 22 | 9
Not completed — Death | 9 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Study terminated by sponsor | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | AZD2811 + Durvalumab | Total
Number analyzed (Participants) | 22 | 9 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (10.4) | 70.4 (7.4) | 65.4 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 18 | 8 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 9 | 29
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 14 | 7 | 21
  White | 8 | 2 | 10
Region of Enrollment [Number; unit: Participants]
  Poland | 3 | 0 | 3
  South Korea | 14 | 7 | 21
  Spain | 3 | 0 | 3
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maintenance Participants Alive and Progression Free (APF12) Per RECIST 1.1 [Efficacy]
Description: 12 month landmark PFS, APF12, where PFS is defined as the time from the first dose of study intervention in the induction phase until objective disease progression (as assessed by the investigator per RECIST v1.1) or death from any cause, whichever comes first.
Time Frame: Up to 12 months
Population: Evaluable population, defined as all participants who entered the maintenance phase and who received at least one dose/have been exposed to any AZD2811 + durvalumab. Only the AZD2811 + durvalumab arm could be evaluable.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
Percentage of patients | NA [NA to NA] — All evaluable patients were either censored or had experienced disease progression (as assessed by the investigator per RECIST v1.1) prior to 12 months post-first-dose of study intervention. Therefore the 12 month PFS landmark estimate was not estimable.

2. Secondary Outcome: Maintenance Participants Alive at 12 Months (OS12), 15 Months (OS15), and 18 Months (OS18)
Description: 12, 15, and 18 month landmarks for Overall Survival (OS) which is defined as the time from the date of first dose of study intervention in the induction phase until death due to any cause, regardless of whether the participant withdraws from study therapy or received another anticancer therapy.
Time Frame: Up to 18 months
Population: Evaluable population, defined as all participants who entered the maintenance phase and who received at least one dose/have been exposed to any AZD2811 + durvalumab. Only the AZD2811 + durvalumab arm could be evaluable.
  The study was terminated early due to the emerging benefit/risk profile of AZD2811. Due to insufficient follow-up at the point of study termination, data were not collected for OS15 and OS18 so these endpoints could not be reported. Only OS12 could be reported.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
Percentage of patients
  OS12 | 33.3 [7.8 to 62.3]
  OS15: number analyzed (Participants) | 0
  OS18: number analyzed (Participants) | 0

3. Secondary Outcome: Maintenance Participants Alive and Progression Free at 6 Months (APF6) and 9 Months (APF9) Using Investigator Assessments According to RECIST 1.1
Description: 6 and 9 month landmark PFS, APF6/APF9, where PFS is defined as the time from the first dose of study intervention in the induction phase until objective disease progression (as assessed by the investigator per RECIST v1.1) or death from any cause, whichever comes first.
Time Frame: Up to 9 months
Population: Evaluable population, defined as all participants who entered the maintenance phase and who received at least one dose/have been exposed to any AZD2811 + durvalumab. The endpoint was not to be collected in patients who did not meet these criteria, so only the AZD2811 + durvalumab arm could be evaluable.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
Percentage of patients
  APF6 | 50.8 [15.7 to 78.1]
  APF9 | 12.7 [0.7 to 42.7]

4. Secondary Outcome: Objective Response Rate (ORR) for All Participants Using Investigator Assessments According to RECIST 1.1
Description: Objective response rate is defined as the percentage of participants with confirmed objective response (CR or PR) per RECIST 1.1. A confirmed response of CR/PR means that a response of CR/PR is recorded at one visit and confirmed by repeat imaging not less than 4 weeks after the visit when the response was first observed with no evidence of progression between the initial and CR/PR confirmation visit.
Time Frame: Up to approximately 10 months
Population: All dosed participants who had measurable disease at baseline. Note that participants were treated for 4 cycles on a Q3W schedule in the induction phase with platinum-based induction therapy (cisplatin or carboplatin plus etoposide) + durvalumab. Participants who had not progressed per RECIST v1.1 at the end of the induction phase and who met maintenance phase eligibility criteria continued into the maintenance phase of the trial and were treated with AZD2811 + durvalumab as maintenance therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Standard of Care | AZD2811 + Durvalumab
Number analyzed (Participants) | 22 | 9
Percentage of patients | 59.1 [36.4 to 79.3] | 77.8 [40.0 to 97.2]

5. Secondary Outcome: Maintenance Participants Progression-free Survival (PFS) Using Investigator Assessments According to RECIST 1.1
Description: Progression-free survival is defined as the time interval from the first dose of study intervention in the induction phase until the date of objective disease progression or death (by any cause, in the absence of progression) regardless of whether the participant withdraws from treatment or received another anticancer therapy prior to progression.
Time Frame: Up to approximately 10 months
Population: Evaluable population, defined as all participants who entered the maintenance phase and who received at least one dose/have been exposed to any AZD2811 + durvalumab. Only the AZD2811+durvlumab arm could be evaluable.
  Due to the early termination of study enrolment, data were not collected up to the intended time frame of 3 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
Months | 6.64 [3.68 to 7.29]

6. Secondary Outcome: Overall Survival (OS) in Maintenance Participants
Description: Overall survival is defined as the time from the date of first dose of study intervention in the induction phase until death due to any cause regardless of whether the subject withdraws from study therapy or receives another anti-cancer therapy.
Time Frame: Up to approximately 13 months
Population: Evaluable population, defined as all participants who entered the maintenance phase and who received at least one dose/have been exposed to any AZD2811 + durvalumab. Only the AZD2811 + durvalumab arm is evaluable.
  Due to the early termination of study enrolment, data were not collected up to the intended time frame of 3 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
Months | 9.99 [4.14 to NA] — Upper confidence limit was not calculable due to an insufficient number of participants with events

7. Secondary Outcome: AZD2811 PK: Pharmacokinetics of AZD2811 and Its Metabolites by Measuring Whole Blood Concentration
Time Frame: Up to Cycle 8 Day 8 (approximately 5 months)
Population: All subjects who received at least one dose of AZD2811 and/or durvalumab with at least one reportable concentration corresponding to the dosed study intervention (reportable means at least one concentration above lower limit of quantification (LLOQ))
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
ng/mL
  AZD2811 Cycle 5 Day 1: Pre-dose: number analyzed (Participants) | 4
  AZD2811 Cycle 5 Day 1: Pre-dose | NA (NA) — All values non reportable as below lower limit of detection
  AZD2811 Cycle 5 Day 1: 2 hours post-dose: number analyzed (Participants) | 4
  AZD2811 Cycle 5 Day 1: 2 hours post-dose | 99264.17 (16.02)
  AZD2811 Cycle 5 Day 3: 2 hours post-dose: number analyzed (Participants) | 5
  AZD2811 Cycle 5 Day 3: 2 hours post-dose | 66764.94 (17.38)
  AZD2811 Cycle 5 Day 8: 2 hours post-dose: number analyzed (Participants) | 5
  AZD2811 Cycle 5 Day 8: 2 hours post-dose | 11024.89 (62.59)
  AZD2811 Cycle 5 Day 15: 2 hours post-dose: number analyzed (Participants) | 4
  AZD2811 Cycle 5 Day 15: 2 hours post-dose | 27.29 (54.45)
  AZD2811 Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 3
  AZD2811 Cycle 6 Day 1: Pre-dose | 18.87 (39.32)
  AZD2811 Cycle 6 Day 1: 2 hours post-dose: number analyzed (Participants) | 6
  AZD2811 Cycle 6 Day 1: 2 hours post-dose | 86706.65 (34.64)
  AZD2811 Cycle 6 Day 8: 2 hours post-dose: number analyzed (Participants) | 7
  AZD2811 Cycle 6 Day 8: 2 hours post-dose | 10827.91 (50.23)
  AZD2811 Cycle 7 Day 1: 2 hours post-dose: number analyzed (Participants) | 4
  AZD2811 Cycle 7 Day 1: 2 hours post-dose | 83625.22 (19.48)
  AZD2811 Cycle 7 Day 8: 2 hours post-dose: number analyzed (Participants) | 3
  AZD2811 Cycle 7 Day 8: 2 hours post-dose | 9004.65 (43.85)
  AZD2811 Cycle 8 Day 1: 2 hours post-dose: number analyzed (Participants) | 3
  AZD2811 Cycle 8 Day 1: 2 hours post-dose | 92287.23 (47.63)
  AZD2811 Cycle 8 Day 8: 2 hours post-dose: number analyzed (Participants) | 3
  AZD2811 Cycle 8 Day 8: 2 hours post-dose | 5839.95 (72.66)
  AZ12102238 Cycle 5 Day 1: Pre-dose: number analyzed (Participants) | 0
  AZ12102238 Cycle 5 Day 1: 2 hours post-dose: number analyzed (Participants) | 3
  AZ12102238 Cycle 5 Day 1: 2 hours post-dose | 3.074 (16.945)
  AZ12102238 Cycle 5 Day 3: 2 hours post-dose: number analyzed (Participants) | 4
  AZ12102238 Cycle 5 Day 3: 2 hours post-dose | 7.379 (16.047)
  AZ12102238 Cycle 5 Day 8: 2 hours post-dose: number analyzed (Participants) | 5
  AZ12102238 Cycle 5 Day 8: 2 hours post-dose | 42.937 (52.690)
  AZ12102238 Cycle 5 Day 15: 2 hours post-dose: number analyzed (Participants) | 4
  AZ12102238 Cycle 5 Day 15: 2 hours post-dose | 18.082 (54.654)
  AZ12102238 Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 5
  AZ12102238 Cycle 6 Day 1: Pre-dose | 8.345 (75.190)
  AZ12102238 Cycle 6 Day 1: 2 hours post-dose: number analyzed (Participants) | 5
  AZ12102238 Cycle 6 Day 1: 2 hours post-dose | 10.099 (62.662)
  AZ12102238 Cycle 6 Day 8: 2 hours post-dose: number analyzed (Participants) | 6
  AZ12102238 Cycle 6 Day 8: 2 hours post-dose | 36.509 (89.757)
  AZ12102238 Cycle 7 Day 1: 2 hours post-dose: number analyzed (Participants) | 4
  AZ12102238 Cycle 7 Day 1: 2 hours post-dose | 9.341 (25.430)
  AZ12102238 Cycle 7 Day 8: 2 hours post-dose: number analyzed (Participants) | 3
  AZ12102238 Cycle 7 Day 8: 2 hours post-dose | 22.117 (16.282)
  AZ12102238 Cycle 8 Day 1: 2 hours post-dose: number analyzed (Participants) | 3
  AZ12102238 Cycle 8 Day 1: 2 hours post-dose | 7.639 (54.423)
  AZ12102238 Cycle 8 Day 8: 2 hours post-dose: number analyzed (Participants) | 3
  AZ12102238 Cycle 8 Day 8: 2 hours post-dose | 28.195 (34.173)

8. Secondary Outcome: EORTC 30: Health Related Quality of Life Based on the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Cancer (QLQ-C30) v3.0.
Description: EORTC QLQ-C30 consists of 30 questions that can be combined to give 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, pain, nausea/vomiting), 6 individual items (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties) and a global measure of health status. QoL issues are assessed using a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) except 2 questions which are between 1 (Very Poor) and 7 (Excellent).
  An outcome variable consisting of a score from 0 to 100 is derived for each scale/item and global health status/QoL. The variable is derived by taking the average of items contributing to a scale or the value of an item and applying a linear transformation to standardize the score, so that scores range from 0 to 100.
  Higher scores on the global health status/QoL and functioning scales indicate better health status/function; higher scores on symptom scales/items represent worse symptoms.
Time Frame: Up to Cycle 10 Day 1, approximately 7 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Standardized score
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
Standardized score
  Physical Functioning: Baseline | 80.00 [60.0 to 93.3]
  Physical Functioning: Cycle 2 Day 1 | 80.00 [26.7 to 100.0]
  Physical Functioning: Cycle 3 Day 1 | 80.00 [40.0 to 100.0]
  Physical Functioning: Cycle 4 Day 1 | 80.00 [40.0 to 93.3]
  Physical Functioning: Cycle 5 Day 1 | 80.00 [60.0 to 100.0]
  Physical Functioning: Cycle 6 Day 1: number analyzed (Participants) | 7
  Physical Functioning: Cycle 6 Day 1 | 80.00 [53.3 to 100.0]
  Physical Functioning: Cycle 7 Day 1: number analyzed (Participants) | 4
  Physical Functioning: Cycle 7 Day 1 | 83.33 [46.7 to 86.7]
  Physical Functioning: Cycle 8 Day 1: number analyzed (Participants) | 2
  Physical Functioning: Cycle 8 Day 1 | 76.67 [73.3 to 80.0]
  Physical Functioning: Cycle 9 Day 1: number analyzed (Participants) | 0
  Physical Functioning: Cycle 10 Day 1: number analyzed (Participants) | 3
  Physical Functioning: Cycle 10 Day 1 | 93.3 [53.3 to 93.3]
  Role functioning: Baseline | 83.33 [66.7 to 100.0]
  Role functioning: Cycle 2 Day 1 | 100.00 [0.0 to 100.0]
  Role functioning: Cycle 3 Day 1 | 83.33 [0.0 to 100.0]
  Role functioning: Cycle 4 Day 1 | 83.33 [0.0 to 100.0]
  Role functioning: Cycle 5 Day 1 | 66.67 [16.7 to 100.0]
  Role functioning: Cycle 6 Day 1: number analyzed (Participants) | 7
  Role functioning: Cycle 6 Day 1 | 83.33 [33.3 to 100.0]
  Role functioning: Cycle 7 Day 1: number analyzed (Participants) | 4
  Role functioning: Cycle 7 Day 1 | 75.00 [33.3 to 100.0]
  Role functioning: Cycle 8 Day 1: number analyzed (Participants) | 2
  Role functioning: Cycle 8 Day 1 | 83.33 [66.7 to 100.0]
  Role functioning: Cycle 9 Day 1: number analyzed (Participants) | 0
  Role functioning: Cycle 10 Day 1: number analyzed (Participants) | 3
  Role functioning: Cycle 10 Day 1 | 100.00 [0.0 to 100.0]
  Cognitive Functioning: Baseline | 83.33 [66.7 to 100.0]
  Cognitive Functioning: Cycle 2 Day 1 | 100.00 [33.3 to 100.0]
  Cognitive Functioning: Cycle 3 Day 1 | 100.00 [33.3 to 100.0]
  Cognitive Functioning: Cycle 4 Day 1 | 100.00 [50.0 to 100.0]
  Cognitive Functioning: Cycle 5 Day 1 | 100.00 [50.0 to 100.0]
  Cognitive Functioning: Cycle 6 Day 1: number analyzed (Participants) | 7
  Cognitive Functioning: Cycle 6 Day 1 | 100.00 [66.7 to 100.0]
  Cognitive Functioning: Cycle 7 Day 1: number analyzed (Participants) | 4
  Cognitive Functioning: Cycle 7 Day 1 | 91.67 [50.0 to 100.0]
  Cognitive Functioning: Cycle 8 Day 1: number analyzed (Participants) | 2
  Cognitive Functioning: Cycle 8 Day 1 | 83.33 [66.7 to 100.0]
  Cognitive Functioning: Cycle 9 Day 1: number analyzed (Participants) | 0
  Cognitive Functioning: Cycle 10 Day 1: number analyzed (Participants) | 3
  Cognitive Functioning: Cycle 10 Day 1 | 66.7 [66.7 to 100.0]
  Emotional Functioning: Baseline | 75.00 [33.3 to 100.0]
  Emotional Functioning: Cycle 2 Day 1 | 91.67 [8.3 to 100.0]
  Emotional Functioning: Cycle 3 Day 1 | 91.67 [41.7 to 100.0]
  Emotional Functioning: Cycle 4 Day 1 | 100.00 [33.3 to 100.0]
  Emotional Functioning: Cycle 5 Day 1 | 100.00 [33.3 to 100.0]
  Emotional Functioning: Cycle 6 Day 1: number analyzed (Participants) | 7
  Emotional Functioning: Cycle 6 Day 1 | 100.0 [33.3 to 100.0]
  Emotional Functioning: Cycle 7 Day 1: number analyzed (Participants) | 4
  Emotional Functioning: Cycle 7 Day 1 | 83.33 [58.3 to 91.7]
  Emotional Functioning: Cycle 8 Day 1: number analyzed (Participants) | 2
  Emotional Functioning: Cycle 8 Day 1 | 91.67 [83.3 to 100.0]
  Emotional Functioning: Cycle 9 Day 1: number analyzed (Participants) | 0
  Emotional Functioning: Cycle 10 Day 1: number analyzed (Participants) | 3
  Emotional Functioning: Cycle 10 Day 1 | 100.00 [50.0 to 100.0]
  Social Functioning: Baseline | 100.00 [66.7 to 100.0]
  Social Functioning: Cycle 2 Day 1 | 83.33 [33.3 to 100.0]
  Social Functioning: Cycle 3 Day 1 | 83.33 [50.0 to 100.0]
  Social Functioning: Cycle 4 Day 1 | 83.33 [16.7 to 100.0]
  Social Functioning: Cycle 5 Day 1 | 83.33 [33.3 to 100.0]
  Social Functioning: Cycle 6 Day 1: number analyzed (Participants) | 7
  Social Functioning: Cycle 6 Day 1 | 83.33 [33.3 to 100.0]
  Social Functioning: Cycle 7 Day 1: number analyzed (Participants) | 4
  Social Functioning: Cycle 7 Day 1 | 83.33 [33.3 to 100.0]
  Social Functioning: Cycle 8 Day 1: number analyzed (Participants) | 2
  Social Functioning: Cycle 8 Day 1 | 91.67 [83.3 to 100.0]
  Social Functioning: Cycle 9 Day 1: number analyzed (Participants) | 0
  Social Functioning: Cycle 10 Day 1: number analyzed (Participants) | 3
  Social Functioning: Cycle 10 Day 1 | 100.00 [50.0 to 100.0]
  Fatigue: Baseline | 22.22 [0.0 to 55.6]
  Fatigue: Cycle 2 Day 1 | 22.22 [0.0 to 100.0]
  Fatigue: Cycle 3 Day 1 | 22.22 [0.0 to 66.7]
  Fatigue: Cycle 4 Day 1 | 33.33 [0.0 to 88.9]
  Fatigue: Cycle 5 Day 1 | 33.33 [0.0 to 77.8]
  Fatigue: Cycle 6 Day 1: number analyzed (Participants) | 7
  Fatigue: Cycle 6 Day 1 | 33.33 [0.0 to 55.6]
  Fatigue: Cycle 7 Day 1: number analyzed (Participants) | 4
  Fatigue: Cycle 7 Day 1 | 27.78 [0.0 to 44.4]
  Fatigue: Cycle 8 Day 1: number analyzed (Participants) | 2
  Fatigue: Cycle 8 Day 1 | 11.11 [0.0 to 22.2]
  Fatigue: Cycle 9 Day 1: number analyzed (Participants) | 0
  Fatigue: Cycle 10 Day 1: number analyzed (Participants) | 3
  Fatigue: Cycle 10 Day 1 | 22.2 [22.2 to 88.9]
  Pain: Baseline | 33.33 [0.0 to 50.0]
  Pain: Cycle 2 Day 1 | 33.33 [0.0 to 100.0]
  Pain: Cycle 3 Day 1 | 16.67 [0.0 to 66.7]
  Pain: Cycle 4 Day 1 | 0.00 [0.0 to 66.7]
  Pain: Cycle 5 Day 1 | 16.67 [0.0 to 66.7]
  Pain: Cycle 6 Day 1: number analyzed (Participants) | 7
  Pain: Cycle 6 Day 1 | 16.67 [0.0 to 33.3]
  Pain: Cycle 7 Day 1: number analyzed (Participants) | 4
  Pain: Cycle 7 Day 1 | 8.33 [0.0 to 16.7]
  Pain: Cycle 8 Day 1: number analyzed (Participants) | 2
  Pain: Cycle 8 Day 1 | 0.00 [0.0 to 0.0]
  Pain: Cycle 9 Day 1: number analyzed (Participants) | 0
  Pain: Cycle 10 Day 1: number analyzed (Participants) | 3
  Pain: Cycle 10 Day 1 | 16.67 [0.0 to 66.7]
  Nausea/Vomiting: Baseline | 0.00 [0.0 to 16.7]
  Nausea/Vomiting: Cycle 2 Day 1 | 0.00 [0.0 to 33.3]
  Nausea/Vomiting: Cycle 3 Day 1 | 0.00 [0.0 to 16.7]
  Nausea/Vomiting: Cycle 4 Day 1 | 0.00 [0.0 to 33.3]
  Nausea/Vomiting: Cycle 5 Day 1 | 0.00 [0.0 to 16.7]
  Nausea/Vomiting: Cycle 6 Day 1: number analyzed (Participants) | 7
  Nausea/Vomiting: Cycle 6 Day 1 | 0.00 [0.0 to 16.7]
  Nausea/Vomiting: Cycle 7 Day 1: number analyzed (Participants) | 4
  Nausea/Vomiting: Cycle 7 Day 1 | 0.00 [0.0 to 16.7]
  Nausea/Vomiting: Cycle 8 Day 1: number analyzed (Participants) | 2
  Nausea/Vomiting: Cycle 8 Day 1 | 0.00 [0.0 to 0.0]
  Nausea/Vomiting: Cycle 9 Day 1: number analyzed (Participants) | 0
  Nausea/Vomiting: Cycle 10 Day 1: number analyzed (Participants) | 3
  Nausea/Vomiting: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Dyspnea: Baseline | 33.33 [0.0 to 66.7]
  Dyspnea: Cycle 2 Day 1 | 33.33 [0.0 to 100.0]
  Dyspnea: Cycle 3 Day 1 | 33.33 [0.0 to 66.7]
  Dyspnea: Cycle 4 Day 1 | 33.33 [0.0 to 66.7]
  Dyspnea: Cycle 5 Day 1 | 33.33 [0.0 to 66.7]
  Dyspnea: Cycle 6 Day 1: number analyzed (Participants) | 7
  Dyspnea: Cycle 6 Day 1 | 33.33 [0.0 to 66.7]
  Dyspnea: Cycle 7 Day 1: number analyzed (Participants) | 4
  Dyspnea: Cycle 7 Day 1 | 33.3 [0.0 to 33.3]
  Dyspnea: Cycle 8 Day 1: number analyzed (Participants) | 2
  Dyspnea: Cycle 8 Day 1 | 50.00 [33.3 to 66.7]
  Dyspnea: Cycle 9 Day 1: number analyzed (Participants) | 0
  Dyspnea: Cycle 10 Day 1: number analyzed (Participants) | 3
  Dyspnea: Cycle 10 Day 1 | 33.33 [0.0 to 66.7]
  Insomnia: Baseline | 0.00 [0.0 to 100.0]
  Insomnia: Cycle 2 Day 1 | 0.00 [0.0 to 100.0]
  Insomnia: Cycle 3 Day 1 | 0.00 [0.0 to 66.7]
  Insomnia: Cycle 4 Day 1 | 0.00 [0.0 to 100.0]
  Insomnia: Cycle 5 Day 1 | 0.00 [0.0 to 66.7]
  Insomnia: Cycle 6 Day 1: number analyzed (Participants) | 7
  Insomnia: Cycle 6 Day 1 | 0.00 [0.0 to 33.3]
  Insomnia: Cycle 7 Day 1: number analyzed (Participants) | 4
  Insomnia: Cycle 7 Day 1 | 0.00 [0.0 to 33.3]
  Insomnia: Cycle 8 Day 1: number analyzed (Participants) | 2
  Insomnia: Cycle 8 Day 1 | 16.67 [0.0 to 33.3]
  Insomnia: Cycle 9 Day 1: number analyzed (Participants) | 0
  Insomnia: Cycle 10 Day 1: number analyzed (Participants) | 3
  Insomnia: Cycle 10 Day 1 | 0.00 [0.0 to 66.7]
  Appetite Loss: Baseline | 33.3 [0.0 to 33.3]
  Appetite Loss: Cycle 2 Day 1 | 33.33 [0.0 to 100.0]
  Appetite Loss: Cycle 3 Day 1 | 33.3 [0.0 to 33.3]
  Appetite Loss: Cycle 4 Day 1 | 33.33 [0.0 to 66.7]
  Appetite Loss: Cycle 5 Day 1 | 0.00 [0.0 to 33.3]
  Appetite Loss: Cycle 6 Day 1: number analyzed (Participants) | 7
  Appetite Loss: Cycle 6 Day 1 | 0.00 [0.0 to 66.7]
  Appetite Loss: Cycle 7 Day 1: number analyzed (Participants) | 4
  Appetite Loss: Cycle 7 Day 1 | 16.67 [0.0 to 33.3]
  Appetite Loss: Cycle 8 Day 1: number analyzed (Participants) | 2
  Appetite Loss: Cycle 8 Day 1 | 16.67 [0.0 to 33.3]
  Appetite Loss: Cycle 9 Day 1: number analyzed (Participants) | 0
  Appetite Loss: Cycle 10 Day 1: number analyzed (Participants) | 3
  Appetite Loss: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Constipation: Baseline | 33.3 [0.0 to 33.3]
  Constipation: Cycle 2 Day 1 | 33.33 [0.0 to 100.0]
  Constipation: Cycle 3 Day 1 | 33.3 [0.0 to 33.3]
  Constipation: Cycle 4 Day 1 | 33.33 [0.0 to 66.7]
  Constipation: Cycle 5 Day 1 | 0.00 [0.0 to 33.3]
  Constipation: Cycle 6 Day 1: number analyzed (Participants) | 7
  Constipation: Cycle 6 Day 1 | 0.00 [0.0 to 66.7]
  Constipation: Cycle 7 Day 1: number analyzed (Participants) | 4
  Constipation: Cycle 7 Day 1 | 16.67 [0.0 to 33.3]
  Constipation: Cycle 8 Day 1: number analyzed (Participants) | 2
  Constipation: Cycle 8 Day 1 | 16.67 [0.0 to 33.3]
  Constipation: Cycle 9 Day 1: number analyzed (Participants) | 0
  Constipation: Cycle 10 Day 1: number analyzed (Participants) | 3
  Constipation: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Diarrhea: Baseline | 0.00 [0.0 to 33.3]
  Diarrhea: Cycle 2 Day 1 | 0.00 [0.0 to 0.0]
  Diarrhea: Cycle 3 Day 1 | 0.00 [0.0 to 33.3]
  Diarrhea: Cycle 4 Day 1 | 0.00 [0.0 to 33.3]
  Diarrhea: Cycle 5 Day 1 | 0.00 [0.0 to 33.3]
  Diarrhea: Cycle 6 Day 1: number analyzed (Participants) | 7
  Diarrhea: Cycle 6 Day 1 | 0.00 [0.0 to 33.3]
  Diarrhea: Cycle 7 Day 1: number analyzed (Participants) | 4
  Diarrhea: Cycle 7 Day 1 | 0.00 [0.0 to 0.0]
  Diarrhea: Cycle 8 Day 1: number analyzed (Participants) | 2
  Diarrhea: Cycle 8 Day 1 | 16.67 [0.0 to 33.3]
  Diarrhea: Cycle 9 Day 1: number analyzed (Participants) | 0
  Diarrhea: Cycle 10 Day 1: number analyzed (Participants) | 3
  Diarrhea: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Financial Difficulties: Baseline | 0.00 [0.0 to 33.3]
  Financial Difficulties: Cycle 2 Day 1 | 0.00 [0.0 to 66.7]
  Financial Difficulties: Cycle 3 Day 1 | 0.00 [0.0 to 100.0]
  Financial Difficulties: Cycle 4 Day 1 | 0.00 [0.0 to 66.7]
  Financial Difficulties: Cycle 5 Day 1 | 0.00 [0.0 to 66.7]
  Financial Difficulties: Cycle 6 Day 1: number analyzed (Participants) | 7
  Financial Difficulties: Cycle 6 Day 1 | 33.33 [0.0 to 100.0]
  Financial Difficulties: Cycle 7 Day 1: number analyzed (Participants) | 4
  Financial Difficulties: Cycle 7 Day 1 | 16.67 [0.0 to 100.0]
  Financial Difficulties: Cycle 8 Day 1: number analyzed (Participants) | 2
  Financial Difficulties: Cycle 8 Day 1 | 0.00 [0.0 to 0.0]
  Financial Difficulties: Cycle 9 Day 1: number analyzed (Participants) | 0
  Financial Difficulties: Cycle 10 Day 1: number analyzed (Participants) | 3
  Financial Difficulties: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Global Health Status: Baseline | 58.33 [33.3 to 91.7]
  Global Health Status: Cycle 2 Day 1 | 66.67 [0.0 to 91.7]
  Global Health Status: Cycle 3 Day 1 | 66.67 [33.3 to 83.3]
  Global Health Status: Cycle 4 Day 1 | 66.67 [25.0 to 100.0]
  Global Health Status: Cycle 5 Day 1 | 66.67 [50.0 to 100.0]
  Global Health Status: Cycle 6 Day 1: number analyzed (Participants) | 7
  Global Health Status: Cycle 6 Day 1 | 83.3 [50.0 to 83.3]
  Global Health Status: Cycle 7 Day 1: number analyzed (Participants) | 4
  Global Health Status: Cycle 7 Day 1 | 70.83 [33.3 to 83.3]
  Global Health Status: Cycle 8 Day 1: number analyzed (Participants) | 2
  Global Health Status: Cycle 8 Day 1 | 66.67 [50.0 to 83.3]
  Global Health Status: Cycle 9 Day 1: number analyzed (Participants) | 0
  Global Health Status: Cycle 10 Day 1: number analyzed (Participants) | 3
  Global Health Status: Cycle 10 Day 1 | 75.00 [33.3 to 83.3]

9. Secondary Outcome: EORTC 13: Lung Cancer Specific Quality of Life Based on the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Lung Cancer (QLQ-LC13) v1.0.
Description: The EORTC QLQ-LC13 is a 13-item questionnaire comprised of 1 symptom scale assessing dysponea, and a series of single questions assessing cough, haemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts, and use of pain medication.
  All items are assessed using a Likert four-point scale (1= not at all to 4 = very much).
  An outcome variable consisting of a score from 0 to 100 is derived for the symptom scale and symptom items according to the EORTC QLQ-LC13 instructions (Fayers et al., 2001). The outcome variable is derived by taking the average of items contributing to a scale or the value of an individual item and applying a linear transformation to standardize the score, so that scores range from 0 to 100.
  Higher scores represent greater symptom severity.
Time Frame: Up to Cycle 10 Day 1, approximately 7 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Standardized score
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
Standardized score
  Alopecia: Baseline | 0.00 [0.0 to 33.3]
  Alopecia: Cycle 2 Day 1 | 66.67 [0.0 to 100.0]
  Alopecia: Cycle 3 Day 1 | 33.33 [0.0 to 100.0]
  Alopecia: Cycle 4 Day 1 | 33.33 [0.0 to 100.0]
  Alopecia: Cycle 5 Day 1 | 0.00 [0.0 to 100.0]
  Alopecia: Cycle 6 Day 1: number analyzed (Participants) | 7
  Alopecia: Cycle 6 Day 1 | 0.00 [0.0 to 100.0]
  Alopecia: Cycle 7 Day 1: number analyzed (Participants) | 4
  Alopecia: Cycle 7 Day 1 | 33.33 [0.0 to 100.0]
  Alopecia: Cycle 8 Day 1: number analyzed (Participants) | 2
  Alopecia: Cycle 8 Day 1 | 16.67 [0.0 to 33.3]
  Alopecia: Cycle 9 Day 1: number analyzed (Participants) | 0
  Alopecia: Cycle 10 Day 1: number analyzed (Participants) | 3
  Alopecia: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Pain in Arm or Shoulder: Baseline | 0.00 [0.0 to 33.3]
  Pain in Arm or Shoulder: Cycle 2 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Arm or Shoulder: Cycle 3 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Arm or Shoulder: Cycle 4 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Arm or Shoulder: Cycle 5 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Arm or Shoulder: Cycle 6 Day 1: number analyzed (Participants) | 7
  Pain in Arm or Shoulder: Cycle 6 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Arm or Shoulder: Cycle 7 Day 1: number analyzed (Participants) | 4
  Pain in Arm or Shoulder: Cycle 7 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Arm or Shoulder: Cycle 8 Day 1: number analyzed (Participants) | 2
  Pain in Arm or Shoulder: Cycle 8 Day 1 | 0.00 [0.0 to 0.0]
  Pain in Arm or Shoulder: Cycle 9 Day 1: number analyzed (Participants) | 0
  Pain in Arm or Shoulder: Cycle 10 Day 1: number analyzed (Participants) | 3
  Pain in Arm or Shoulder: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Pain in Chest: Baseline | 33.33 [0.0 to 66.7]
  Pain in Chest: Cycle 2 Day 1 | 33.33 [0.0 to 66.7]
  Pain in Chest: Cycle 3 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Chest: Cycle 4 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Chest: Cycle 5 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Chest: Cycle 6 Day 1: number analyzed (Participants) | 7
  Pain in Chest: Cycle 6 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Chest: Cycle 7 Day 1: number analyzed (Participants) | 4
  Pain in Chest: Cycle 7 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Chest: Cycle 8 Day 1: number analyzed (Participants) | 2
  Pain in Chest: Cycle 8 Day 1 | 33.3 [33.3 to 33.3]
  Pain in Chest: Cycle 9 Day 1: number analyzed (Participants) | 0
  Pain in Chest: Cycle 10 Day 1: number analyzed (Participants) | 3
  Pain in Chest: Cycle 10 Day 1 | 0.00 [0.0 to 33.3]
  Coughing: Baseline | 33.33 [33.3 to 66.7]
  Coughing: Cycle 2 Day 1 | 33.33 [0.0 to 66.7]
  Coughing: Cycle 3 Day 1 | 0.00 [0.0 to 66.7]
  Coughing: Cycle 4 Day 1 | 0.00 [0.0 to 66.7]
  Coughing: Cycle 5 Day 1 | 0.00 [0.0 to 66.7]
  Coughing: Cycle 6 Day 1: number analyzed (Participants) | 7
  Coughing: Cycle 6 Day 1 | 33.33 [0.0 to 66.7]
  Coughing: Cycle 7 Day 1: number analyzed (Participants) | 4
  Coughing: Cycle 7 Day 1 | 33.33 [0.0 to 66.7]
  Coughing: Cycle 8 Day 1: number analyzed (Participants) | 2
  Coughing: Cycle 8 Day 1 | 33.33 [0.0 to 66.7]
  Coughing: Cycle 9 Day 1: number analyzed (Participants) | 0
  Coughing: Cycle 10 Day 1: number analyzed (Participants) | 3
  Coughing: Cycle 10 Day 1 | 0.00 [0.0 to 66.7]
  Dysphagia: Baseline | 0.00 [0.0 to 33.3]
  Dysphagia: Cycle 2 Day 1 | 0.00 [0.0 to 100.0]
  Dysphagia: Cycle 3 Day 1 | 0.00 [0.0 to 0.0]
  Dysphagia: Cycle 4 Day 1 | 0.00 [0.0 to 0.0]
  Dysphagia: Cycle 5 Day 1 | 0.00 [0.0 to 33.3]
  Dysphagia: Cycle 6 Day 1: number analyzed (Participants) | 7
  Dysphagia: Cycle 6 Day 1 | 0.00 [0.0 to 66.7]
  Dysphagia: Cycle 7 Day 1: number analyzed (Participants) | 4
  Dysphagia: Cycle 7 Day 1 | 0.00 [0.0 to 33.3]
  Dysphagia: Cycle 8 Day 1: number analyzed (Participants) | 2
  Dysphagia: Cycle 8 Day 1 | 0.00 [0.0 to 0.0]
  Dysphagia: Cycle 9 Day 1: number analyzed (Participants) | 0
  Dysphagia: Cycle 10 Day 1: number analyzed (Participants) | 3
  Dysphagia: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Dyspnea: Baseline | 22.22 [0.0 to 55.6]
  Dyspnea: Cycle 2 Day 1 | 22.22 [0.0 to 66.7]
  Dyspnea: Cycle 3 Day 1 | 22.22 [11.1 to 66.7]
  Dyspnea: Cycle 4 Day 1 | 22.22 [11.1 to 66.7]
  Dyspnea: Cycle 5 Day 1 | 33.33 [0.0 to 66.7]
  Dyspnea: Cycle 6 Day 1: number analyzed (Participants) | 7
  Dyspnea: Cycle 6 Day 1 | 33.33 [0.0 to 66.7]
  Dyspnea: Cycle 7 Day 1: number analyzed (Participants) | 4
  Dyspnea: Cycle 7 Day 1 | 22.22 [0.0 to 33.3]
  Dyspnea: Cycle 8 Day 1: number analyzed (Participants) | 2
  Dyspnea: Cycle 8 Day 1 | 27.78 [22.2 to 33.3]
  Dyspnea: Cycle 9 Day 1: number analyzed (Participants) | 0
  Dyspnea: Cycle 10 Day 1: number analyzed (Participants) | 3
  Dyspnea: Cycle 10 Day 1 | 44.4 [22.2 to 44.4]
  Hemoptysis: Baseline | 0.00 [0.0 to 33.3]
  Hemoptysis: Cycle 2 Day 1 | 0.00 [0.0 to 0.0]
  Hemoptysis: Cycle 3 Day 1 | 0.00 [0.0 to 0.0]
  Hemoptysis: Cycle 4 Day 1 | 0.00 [0.0 to 0.0]
  Hemoptysis: Cycle 5 Day 1 | 0.00 [0.0 to 0.0]
  Hemoptysis: Cycle 6 Day 1: number analyzed (Participants) | 7
  Hemoptysis: Cycle 6 Day 1 | 0.00 [0.0 to 33.3]
  Hemoptysis: Cycle 7 Day 1: number analyzed (Participants) | 4
  Hemoptysis: Cycle 7 Day 1 | 0.00 [0.0 to 0.0]
  Hemoptysis: Cycle 8 Day 1: number analyzed (Participants) | 2
  Hemoptysis: Cycle 8 Day 1 | 0.00 [0.0 to 0.0]
  Hemoptysis: Cycle 9 Day 1: number analyzed (Participants) | 0
  Hemoptysis: Cycle 10 Day 1: number analyzed (Participants) | 3
  Hemoptysis: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]
  Pain in Other Parts: Baseline | 33.33 [0.0 to 66.7]
  Pain in Other Parts: Cycle 2 Day 1 | 33.33 [0.0 to 100.0]
  Pain in Other Parts: Cycle 3 Day 1 | 33.33 [0.0 to 100.0]
  Pain in Other Parts: Cycle 4 Day 1 | 0.00 [0.0 to 100.0]
  Pain in Other Parts: Cycle 5 Day 1 | 0.00 [0.0 to 100.0]
  Pain in Other Parts: Cycle 6 Day 1: number analyzed (Participants) | 7
  Pain in Other Parts: Cycle 6 Day 1 | 0.00 [0.0 to 33.3]
  Pain in Other Parts: Cycle 7 Day 1: number analyzed (Participants) | 4
  Pain in Other Parts: Cycle 7 Day 1 | 16.67 [0.0 to 33.3]
  Pain in Other Parts: Cycle 8 Day 1: number analyzed (Participants) | 2
  Pain in Other Parts: Cycle 8 Day 1 | 16.67 [0.0 to 33.3]
  Pain in Other Parts: Cycle 9 Day 1: number analyzed (Participants) | 0
  Pain in Other Parts: Cycle 10 Day 1: number analyzed (Participants) | 3
  Pain in Other Parts: Cycle 10 Day 1 | 33.3 [33.3 to 33.3]
  Peripheral Neuropathy: Baseline | 0.00 [0.0 to 33.3]
  Peripheral Neuropathy: Cycle 2 Day 1 | 33.33 [0.0 to 100.0]
  Peripheral Neuropathy: Cycle 3 Day 1 | 0.00 [0.0 to 33.3]
  Peripheral Neuropathy: Cycle 4 Day 1 | 0.00 [0.0 to 100.0]
  Peripheral Neuropathy: Cycle 5 Day 1 | 0.00 [0.0 to 66.7]
  Peripheral Neuropathy: Cycle 6 Day 1: number analyzed (Participants) | 7
  Peripheral Neuropathy: Cycle 6 Day 1 | 0.00 [0.0 to 33.3]
  Peripheral Neuropathy: Cycle 7 Day 1: number analyzed (Participants) | 4
  Peripheral Neuropathy: Cycle 7 Day 1 | 0.00 [0.0 to 33.3]
  Peripheral Neuropathy: Cycle 8 Day 1: number analyzed (Participants) | 2
  Peripheral Neuropathy: Cycle 8 Day 1 | 0.00 [0.0 to 0.0]
  Peripheral Neuropathy: Cycle 9 Day 1: number analyzed (Participants) | 0
  Peripheral Neuropathy: Cycle 10 Day 1: number analyzed (Participants) | 3
  Peripheral Neuropathy: Cycle 10 Day 1 | 33.33 [0.0 to 66.7]
  Sore Mouth: Baseline | 0.00 [0.0 to 33.3]
  Sore Mouth: Cycle 2 Day 1 | 0.00 [0.0 to 100.0]
  Sore Mouth: Cycle 3 Day 1 | 0.00 [0.0 to 0.0]
  Sore Mouth: Cycle 4 Day 1 | 0.00 [0.0 to 0.0]
  Sore Mouth: Cycle 5 Day 1 | 0.00 [0.0 to 0.0]
  Sore Mouth: Cycle 6 Day 1: number analyzed (Participants) | 7
  Sore Mouth: Cycle 6 Day 1 | 0.00 [0.0 to 33.3]
  Sore Mouth: Cycle 7 Day 1: number analyzed (Participants) | 4
  Sore Mouth: Cycle 7 Day 1 | 0.00 [0.0 to 0.0]
  Sore Mouth: Cycle 8 Day 1: number analyzed (Participants) | 2
  Sore Mouth: Cycle 8 Day 1 | 0.00 [0.0 to 0.0]
  Sore Mouth: Cycle 9 Day 1: number analyzed (Participants) | 0
  Sore Mouth: Cycle 10 Day 1: number analyzed (Participants) | 3
  Sore Mouth: Cycle 10 Day 1 | 0.00 [0.0 to 0.0]

10. Secondary Outcome: EORTC 13: Lung Cancer Specific Quality of Life Based on the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Lung Cancer (QLQ-LC13) v1.0. Use of Pain Medication (Yes/No)
Description: The EORTC QLQ-LC13 is a 13-item questionnaire comprised of 1 symptom scale assessing dysponea, and a series of single questions assessing cough, haemoptysis, sore mouth, dysphagis, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts, and use of pain medication. Use of pain medication is collected as a Yes/No response.
Time Frame: Up to Cycle 10 Day 1, approximately 7 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2811 + Durvalumab
Number analyzed (Participants) | 9
Participants
  Use of Pain Medication: Baseline: Yes | 3
  Use of Pain Medication: Baseline: No | 6
  Use of Pain Medication: Cycle 2 Day 1: Yes | 8
  Use of Pain Medication: Cycle 2 Day 1: No | 1
  Use of Pain Medication: Cycle 3 Day 1: Yes | 5
  Use of Pain Medication: Cycle 3 Day 1: No | 4
  Use of Pain Medication: Cycle 4 Day 1: Yes | 4
  Use of Pain Medication: Cycle 4 Day 1: No | 5
  Use of Pain Medication: Cycle 5 Day 1: Yes | 4
  Use of Pain Medication: Cycle 5 Day 1: No | 5
  Use of Pain Medication: Cycle 6 Day 1: number analyzed (Participants) | 7
  Use of Pain Medication: Cycle 6 Day 1: Yes | 2
  Use of Pain Medication: Cycle 6 Day 1: No | 5
  Use of Pain Medication: Cycle 7 Day 1: number analyzed (Participants) | 4
  Use of Pain Medication: Cycle 7 Day 1: Yes | 1
  Use of Pain Medication: Cycle 7 Day 1: No | 3
  Use of Pain Medication: Cycle 8 Day 1: number analyzed (Participants) | 2
  Use of Pain Medication: Cycle 8 Day 1: Yes | 1
  Use of Pain Medication: Cycle 8 Day 1: No | 1
  Use of Pain Medication: Cycle 9 Day 1: number analyzed (Participants) | 0
  Use of Pain Medication: Cycle 10 Day 1: number analyzed (Participants) | 3
  Use of Pain Medication: Cycle 10 Day 1: Yes | 3
  Use of Pain Medication: Cycle 10 Day 1: No | 0

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events (TEAEs) were collected up to the final analysis DCO, maximum of approximately 16 months.
Description: TEAEs included those from first administration of study treatment up to and including 90 days after last dose of study treatment or up to date of initiation of the first subsequent anticancer therapy (whichever occurred first).
Groups:
- Induction Phase SoC; Induction Phase AZD2811 + Durva; Maintenance Phase SoC; Maintenance Phase AZD2811 + Durva: Description (Arm-group)
Arm/Group | Induction Phase SoC | Induction Phase AZD2811 + Durva | Maintenance Phase SoC | Maintenance Phase AZD2811 + Durva
All-Cause Mortality (participants affected / at risk) | 6/22 | 0/9 | 3/13 | 6/9
Serious Adverse Events (participants affected / at risk) | 6/22 | 3/9 | 0/13 | 6/9
Other Adverse Events (participants affected / at risk) | 21/22 | 9/9 | 6/13 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Phase SoC (N=22) | Induction Phase AZD2811 + Durva (N=9) | Maintenance Phase SoC (N=13) | Maintenance Phase AZD2811 + Durva (N=9)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Phase SoC (N=22) | Induction Phase AZD2811 + Durva (N=9) | Maintenance Phase SoC (N=13) | Maintenance Phase AZD2811 + Durva (N=9)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 8 (10) | 7 (9) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood chloride decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 11 (28) | 7 (19) | 1 (1) | 7 (10)
Platelet count decreased (Investigations) | 2 (3) | 2 (3) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (11) | 1 (2) | 0 (0) | 0 (0)
Thyroid function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (6) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (8) | 4 (7) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrolment to Study D6132C00001 was terminated prior to completion of the study due to the evolving benefit-risk profile of AZD2811 not supporting further development for the first-line treatment of patients with extensive stage small-cell lung cancer (ES-SCLC). Due to the early termination of the study, only 9 participants (of the planned 80 participants) received maintenance treatment with AZD2811 in combination with durvalumab and data collection for these participants was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04745689/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT04745689/SAP_001.pdf